CLINICAL TRIAL: NCT01159847
Title: Protective Effects of Sitagliptin on β Cell Function in Patients With Adult-onset Latent Autoimmune Diabetes (LADA)
Acronym: DPP-ⅣLADA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Foundation for the Study of Diabetes (Other)
Collaborators: Chinese Medical Association (Network); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director, Department of Endocrinology, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFSD DPP-Ⅳ LADA
Record Dates: First submitted 2010-05-05; First posted 2010-07-12 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes
Keywords: sitagliptin; LADA; C-Peptide; Flow Cytometry; ELISPOT
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Patients will receive insulin therapy with sitagliptin.
  Interventions: Drug: sitagliptin; Drug: Insulin
- Insulin (Active Comparator): Patients will receive insulin therapy without sitagliptin.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: sitagliptin — sitagliptin tablet,100 mg p.o. qd,2 year
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Insulin

SUMMARY:
The aim of this study is to investigate the protective effects of sitagliptin on β cell function in patients with adult-onset latent autoimmune diabetes (LADA) and its mechanisms.

DETAILED DESCRIPTION:
Adult-onset latent autoimmune diabetes (LADA), etiologically belongs to type 1 diabetes (T1D), is characterized by the presence of islet autoantibodies, such as islet cell antibody (ICA) and glutamic acid decarboxylase antibody (GADA), and is prone to develop β-cell failure. The goals of treatment for LADA are suppression of autoimmune β cell destruction, preservation of islet function and prevention of diabetic complications. Recently two classes of compounds have been approved by the FDA as type 2 diabetes (T2D) therapeutics: the glucagon-like peptide-1 (GLP-1) receptor agonist (incretin mimetic) exenatide (Byetta) and the dipeptidyl peptidase IV (DPP-IV) inhibitor sitagliptin (Januvia) and vildagliptin (Galvus). They have been shown to reduce HbA1c, fasting glucose and to improve β cell function in T2D patients, as a mono-therapy or in combination with metformin or thiazolidinediones. Besides, in vitro studies showed incretin-based therapy can stimulate β-cell proliferation and survival, increase β cell insulin content and inhibit apoptosis. Moreover, several short-term pilot studies suggest GLP-1 may also have the potential for treating T1D. Several findings suggest that Ex-4 may also act as a regulator of the immune response in addition to its potential effects on β cell proliferation. Therefore, we hypothesized DPP-IV inhibitors might provide therapeutic advantages in T1D though no study has been reported. Besides the β cell function, another important target is insulin sensitivity. As for DPP-IV inhibitor, clinical trials demonstrated their beneficial effects on insulin sensitivity in subjects with T2D and impaired fasting glucose (IFG) and in diabetic rat model. We'd like to further explore the possible effect of sitagliptin on insulin sensitivity in LADA patients by homeostasis model assessment for insulin resistance (HOMA-IR) index and euglycemic clamp technique. In addition, the systemic inflammation associated with a wide array of plasma proteins and pro-inflammatory cytokines (i.e., C reactive protein (CRP), tumor necrosis factor-α (TNF-α), interleukin-6) play an additional role in the pathogenesis of insulin resistance in diabetes. It will be of interest to investigate the adipokines and proinflammatory cytokines after the sitagliptin therapy in the study. Hence, we aim to explore the effects of sitagliptin plus insulin on β cell function, insulin sensitivity, pro-inflammatory cytokines and immune regulation including Teff and Treg frequency, and function in patients with LADA.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes diagnosed according to the report of WHO in 1999.
2. Age at onset between 25~70 years.
3. Disease duration of less than 3 year.
4. No ketoacidosis within the first 6 months after diagnosis of diabetes.
5. GADA positive twice within one month.
6. Fasting C-peptide (FCP) level of 0.2 nmol/L or more.

Exclusion Criteria:

1. Insulin requirements more than 0.8 units/kg/day.
2. Evidence of chronic infection or acute infection affected blood glucose control within 4 weeks prior to visit 1.
3. History of any malignancy.
4. Pregnancy, breastfeeding or planned pregnancy within two years.
5. Secondary diabetes.
6. Congestive heart failure requiring pharmacologic treatment.
7. Renal disease or renal dysfunction or diabetic nephropathy suggested by serum creatinine levels≥1.5 mg/dL (132μmol/L) for males and ≥1.4mg/dL (123μmol/L) for females or abnormal creatinine clearance at Visit 1.
8. Concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The effects of sitagliptin on β cell function and insulin sensitivity of LADA patients | 2 years
  1. The assessment of the change of β cell function in patients with LADA treated with sitagliptin plus insulin by the standardized mixed meal stimulation test and insulin sensitivity by HOMA-IR.
  2. The assessment of the change of insulin sensitivity in LADA patients by sequential insulin infusion with the euglycemic glucose clamp technique.

SECONDARY OUTCOMES:
The possible immunomodulatory effects of sitagliptin on LADA patients | 2 years
  The change of the frequency of pathogenic Teff (CD4+Th1, Th2, Th17 and CD8+) cells and CD4+CD25+Foxp3+Treg cells before and after sitagliptin treatment in LADA patients.
The possible immunomodulatory effects of sitagliptin on LADA patients | 2 years
  Effect of sitagliptin on cytokine production of Teff and Treg cells before and after sitagliptin treatment in LADA patients.
The possible immunomodulatory effects of sitagliptin on LADA patients | 2 years
  Effect of sitagliptin on Foxp3 mRNA expression of Treg cells and RORγT mRNA expression of Th17 cells before and after sitagliptin treatment in LADA patients.
The possible immunomodulatory effects of sitagliptin on LADA patients | 2 years
  The comparison of glutamic acid decarboxylase 65 (GAD65) reactive interferon-γ-Th1, IL-4-Th2, IL-17-Th17 and IL-10-Treg cells detected by enzyme-linked immunospot (ELISPOT) before and after sitagliptin treatment in LADA patients.
The possible immunomodulatory effects of sitagliptin on LADA patients | 2 years
  The change of the adiponectin, IL-6, IL-17 and CRP etc. before and after the sitagliptin treatment in LADA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, M.D., Ph.D., Principal Investigator — Diabetes Center, Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, China
Locations (1):
- Diabetes Center, Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Tuomi T, Groop LC, Zimmet PZ, Rowley MJ, Knowles W, Mackay IR. Antibodies to glutamic acid decarboxylase reveal latent autoimmune diabetes mellitus in adults with a non-insulin-dependent onset of disease. Diabetes. 1993 Feb;42(2):359-62. doi: 10.2337/diab.42.2.359. PMID 8425674
- [Background] Dupre J. Glycaemic effects of incretins in Type 1 diabetes mellitus: a concise review, with emphasis on studies in humans. Regul Pept. 2005 Jun 15;128(2):149-57. doi: 10.1016/j.regpep.2004.06.003. PMID 15780434
- [Background] Dupre J, Behme MT, Hramiak IM, McFarlane P, Williamson MP, Zabel P, McDonald TJ. Glucagon-like peptide I reduces postprandial glycemic excursions in IDDM. Diabetes. 1995 Jun;44(6):626-30. doi: 10.2337/diab.44.6.626. PMID 7789625
- [Background] Behme MT, Dupre J, McDonald TJ. Glucagon-like peptide 1 improved glycemic control in type 1 diabetes. BMC Endocr Disord. 2003 Apr 10;3(1):3. doi: 10.1186/1472-6823-3-3. PMID 12697069
- [Background] Creutzfeldt WO, Kleine N, Willms B, Orskov C, Holst JJ, Nauck MA. Glucagonostatic actions and reduction of fasting hyperglycemia by exogenous glucagon-like peptide I(7-36) amide in type I diabetic patients. Diabetes Care. 1996 Jun;19(6):580-6. doi: 10.2337/diacare.19.6.580. PMID 8725855
- [Background] Zhang J, Tokui Y, Yamagata K, Kozawa J, Sayama K, Iwahashi H, Okita K, Miuchi M, Konya H, Hamaguchi T, Namba M, Shimomura I, Miyagawa JI. Continuous stimulation of human glucagon-like peptide-1 (7-36) amide in a mouse model (NOD) delays onset of autoimmune type 1 diabetes. Diabetologia. 2007 Sep;50(9):1900-1909. doi: 10.1007/s00125-007-0737-6. Epub 2007 Jul 14. PMID 17632702
- [Background] Pospisilik JA, Martin J, Doty T, Ehses JA, Pamir N, Lynn FC, Piteau S, Demuth HU, McIntosh CH, Pederson RA. Dipeptidyl peptidase IV inhibitor treatment stimulates beta-cell survival and islet neogenesis in streptozotocin-induced diabetic rats. Diabetes. 2003 Mar;52(3):741-50. doi: 10.2337/diabetes.52.3.741. PMID 12606516
- [Background] Pospisilik JA, Ehses JA, Doty T, McIntosh CH, Demuth HU, Pederson RA. Dipeptidyl peptidase IV inhibition in animal models of diabetes. Adv Exp Med Biol. 2003;524:281-91. doi: 10.1007/0-306-47920-6_34. No abstract available. PMID 12675250
- [Background] Kim SJ, Nian C, Doudet DJ, McIntosh CH. Inhibition of dipeptidyl peptidase IV with sitagliptin (MK0431) prolongs islet graft survival in streptozotocin-induced diabetic mice. Diabetes. 2008 May;57(5):1331-9. doi: 10.2337/db07-1639. Epub 2008 Feb 25. PMID 18299314
- [Background] Flentke GR, Munoz E, Huber BT, Plaut AG, Kettner CA, Bachovchin WW. Inhibition of dipeptidyl aminopeptidase IV (DP-IV) by Xaa-boroPro dipeptides and use of these inhibitors to examine the role of DP-IV in T-cell function. Proc Natl Acad Sci U S A. 1991 Feb 15;88(4):1556-9. doi: 10.1073/pnas.88.4.1556. PMID 1671716
- [Background] Reinhold D, Bank U, Buhling F, Lendeckel U, Faust J, Neubert K, Ansorge S. Inhibitors of dipeptidyl peptidase IV induce secretion of transforming growth factor-beta 1 in PWM-stimulated PBMC and T cells. Immunology. 1997 Jul;91(3):354-60. doi: 10.1046/j.1365-2567.1997.d01-2258.x. PMID 9301523
- [Background] Kahne T, Neubert K, Faust J, Ansorge S. Early phosphorylation events induced by DPIV/CD26-specific inhibitors. Cell Immunol. 1998 Oct 10;189(1):60-6. doi: 10.1006/cimm.1998.1355. PMID 9758695
- [Background] Yang Z, Zhou Z, Huang G, Ling H, Yan X, Peng J, Li X. The CD4(+) regulatory T-cells is decreased in adults with latent autoimmune diabetes. Diabetes Res Clin Pract. 2007 Apr;76(1):126-31. doi: 10.1016/j.diabres.2006.08.013. Epub 2006 Sep 26. PMID 17005288
- [Background] Xue S, Wasserfall CH, Parker M, Brusko TM, McGrail S, McGrail K, Moore M, Campbell-Thompson M, Schatz DA, Atkinson MA, Haller MJ. Exendin-4 therapy in NOD mice with new-onset diabetes increases regulatory T cell frequency. Ann N Y Acad Sci. 2008 Dec;1150:152-6. doi: 10.1196/annals.1447.049. PMID 19120286
- [Background] Utzschneider KM, Tong J, Montgomery B, Udayasankar J, Gerchman F, Marcovina SM, Watson CE, Ligueros-Saylan MA, Foley JE, Holst JJ, Deacon CF, Kahn SE. The dipeptidyl peptidase-4 inhibitor vildagliptin improves beta-cell function and insulin sensitivity in subjects with impaired fasting glucose. Diabetes Care. 2008 Jan;31(1):108-13. doi: 10.2337/dc07-1441. Epub 2007 Oct 1. PMID 17909087
- [Background] Ahren B, Pacini G, Foley JE, Schweizer A. Improved meal-related beta-cell function and insulin sensitivity by the dipeptidyl peptidase-IV inhibitor vildagliptin in metformin-treated patients with type 2 diabetes over 1 year. Diabetes Care. 2005 Aug;28(8):1936-40. doi: 10.2337/diacare.28.8.1936. PMID 16043735
- [Background] Orskov L, Holst JJ, Moller J, Orskov C, Moller N, Alberti KG, Schmitz O. GLP-1 does not not acutely affect insulin sensitivity in healthy man. Diabetologia. 1996 Oct;39(10):1227-32. doi: 10.1007/BF02658511. PMID 8897012
- [Background] Ahren B, Larsson H, Holst JJ. Effects of glucagon-like peptide-1 on islet function and insulin sensitivity in noninsulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1997 Feb;82(2):473-8. doi: 10.1210/jcem.82.2.3728. PMID 9024239
- [Background] Zander M, Madsbad S, Madsen JL, Holst JJ. Effect of 6-week course of glucagon-like peptide 1 on glycaemic control, insulin sensitivity, and beta-cell function in type 2 diabetes: a parallel-group study. Lancet. 2002 Mar 9;359(9309):824-30. doi: 10.1016/S0140-6736(02)07952-7. PMID 11897280
- [Background] Pospisilik JA, Stafford SG, Demuth HU, McIntosh CH, Pederson RA. Long-term treatment with dipeptidyl peptidase IV inhibitor improves hepatic and peripheral insulin sensitivity in the VDF Zucker rat: a euglycemic-hyperinsulinemic clamp study. Diabetes. 2002 Sep;51(9):2677-83. doi: 10.2337/diabetes.51.9.2677. PMID 12196458
- [Background] Pietropaolo M, Barinas-Mitchell E, Kuller LH. The heterogeneity of diabetes: unraveling a dispute: is systemic inflammation related to islet autoimmunity? Diabetes. 2007 May;56(5):1189-97. doi: 10.2337/db06-0880. Epub 2007 Feb 23. PMID 17322478
- [Background] Viswanathan P, Chaudhuri A, Bhatia R, Al-Atrash F, Mohanty P, Dandona P. Exenatide therapy in obese patients with type 2 diabetes mellitus treated with insulin. Endocr Pract. 2007 Sep;13(5):444-50. doi: 10.4158/EP.13.5.444. PMID 17872344
- [Background] Duttaroy A, Voelker F, Merriam LQ, et al. The DPP-4 inhibitor Vildagliptin increases pancreatic β-cell neogenesis and decreases apoptosis. Diabetes, 2005; 54 (Suppl. 1): A141.
- [Background] Yang ZF, Zhou ZG, Tang WL, Huang G, Peng J, Li X, He L. [Decrease of FOXP3 mRNA in CD4+ T cells in latent autoimmune diabetes in adult]. Zhonghua Yi Xue Za Zhi. 2006 Sep 26;86(36):2533-6. Chinese. PMID 17198560
- [Background] Korom S, De Meester I, Stadlbauer TH, Chandraker A, Schaub M, Sayegh MH, Belyaev A, Haemers A, Scharpe S, Kupiec-Weglinski JW. Inhibition of CD26/dipeptidyl peptidase IV activity in vivo prolongs cardiac allograft survival in rat recipients. Transplantation. 1997 May 27;63(10):1495-500. doi: 10.1097/00007890-199705270-00021. PMID 9175816
- [Derived] Yang L, Liang H, Liu X, Wang X, Cheng Y, Zhao Y, Liu L, Huang G, Wang X, Zhou Z. Islet Function and Insulin Sensitivity in Latent Autoimmune Diabetes in Adults Taking Sitagliptin: A Randomized Trial. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1529-e1541. doi: 10.1210/clinem/dgab026. PMID 33475138
- [Derived] Wang X, Yang L, Cheng Y, Liang H, Hu J, Zheng P, Huang G, Zhou Z. Downregulation of T-Cell Transcription Factors in Adult Latent Autoimmune Diabetes with High-Titer Glutamic Acid Decaroxylase Antibody. Diabetes Ther. 2019 Jun;10(3):917-927. doi: 10.1007/s13300-019-0594-6. Epub 2019 Mar 20. PMID 30895467
- [Derived] Zhao Y, Yang L, Xiang Y, Liu L, Huang G, Long Z, Li X, Leslie RD, Wang X, Zhou Z. Dipeptidyl peptidase 4 inhibitor sitagliptin maintains beta-cell function in patients with recent-onset latent autoimmune diabetes in adults: one year prospective study. J Clin Endocrinol Metab. 2014 May;99(5):E876-80. doi: 10.1210/jc.2013-3633. Epub 2014 Jan 16. PMID 24432999